CLINICAL TRIAL: NCT04184479
Title: Placebo-Controlled, Randomized Weight Loss InterventionTrial in Subjects With Overweight or Obesity in Primary Health Care
Brief Title: Effect of the LEVAmethod by Bertz et al © in Subjects With Overweight or Obesity in Primary Health Care.
Acronym: LEVA-POP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEVA-POP
Record Dates: First submitted 2019-11-24; First posted 2019-12-03 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Overweight and Obesity
Keywords: overweight; randomized controlled trial; obesity; weight loss; weight loss maintenance
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-LEVAmetoden by Bertz et al (Active Comparator): Individual dietary advices for weight loss, based on the participants' food record of 4 consecutive days aimed to achieve an energy intake reduction of 500 kcal/d with a nutrient composition according to the Nordic Nutrition Recommendations. Follow up visits after 3 months, 1 year and 2 years after baseline. Follow up by electronic platform every other week until 3 months after baseline and each month after 3 months until 1 year after baseline.
  Interventions: Behavioral: LEVAmethod by Bertz et al
- B-Ordinary treatment (Placebo Comparator): Dietary advices for weight loss aimed to achieve calorie restriction. Follow up visits after 3 months, 1 year and 2 years after baseline. Additional visits, up to 4 times in the first year after baseline.
  Interventions: Behavioral: LEVAmethod by Bertz et al

INTERVENTIONS:
Behavioral: LEVAmethod by Bertz et al — Ordinary treatment
  Other Names: Ordinary treatment

SUMMARY:
This study evaluates weight loss effect of the method LEVA by Bertz et al in subjects with overweight or obesity that are remitted to Primärvårdens Dietistenhet.

DETAILED DESCRIPTION:
The method "Lifestyle at Effective Weight Loss During Breastfeeding" (LEVA method by Bertz et al) has been scientifically studied to provide sustainable weight loss for women with overweight or obesity after childbirth. Primary health care centers in Västra Götalandsregionen treat adult patients with overweight and obesity. If the LEVA method by Bertz et el also produces weight loss to other patient groups than women post partum, the method could be used as a treatment alternative.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27 ≤ 35
* age 18-75 år

Exclusion Criteria:

* difficulty understanding Swedish, spoken or read
* does not manage/want to handle digital Tools
* the remittance was addressed to Primärvårdens Dietistenhet at wrong premises and the patient should be treated elsewhere.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change of weight between intervention group and placebo | From baseline and 12 weeks
  Weight in kg measured at visits
Change of weight between intervention group and placebo | From baseline and 1 year
  Weight in kg measured at visits
Change of weight between intervention group and placebo | From baseline and 2 year
  Weight in kg measured at visits

SECONDARY OUTCOMES:
Gender differences in weight loss results | From baseline to 12 weeks
  weight in kg measured at visits in relation to gender
Gender differences in weight loss results | From baseline to 1 year
  weight in kg measured at visits in relation to gender
Gender differences in weight loss results | From baseline to 2 year
  weight in kg measured at visits in relation to gender
Age differences in weight loss results | From baseline to 12 weeks
  Weight in kg measured at visits in relation to age
Age differences in weight loss results | From baseline to 1 years
  Weight in kg measured at visits in relation to age
Age differences in weight loss results | From baseline to 2 years
  Weight in kg measured at visits in relation to age
Weight loss result in relation to pre-treatment BMI | From baseline to 12 weeks
  Weight in kg measured at visits in relation to pre-treatment BMI
Weight loss result in relation to pre-treatment BMI | From baseline to 1 year
  Weight in kg measured at visits in relation to pre-treatment BMI
Weight loss result in relation to pre-treatment BMI | From baseline to 2 year
  Weight in kg measured at visits in relation to pre-treatment BMI
Cost-effectiveness of LEVA method by Bertz et al | From baseline to 12 weeks
  Calculation of cost-effectiveness by the method of monetary net benefit
Cost-effectiveness of LEVA method by Bertz et al | From baseline to 1 year
  Calculation of cost-effectiveness by the method of monetary net benefit
Cost-effectiveness of LEVA method by Bertz et al | From baseline to 2 year
  Calculation of cost-effectiveness by the method of monetary net benefit

CONTACTS AND LOCATIONS:
Overall Officials: Else Johansson, Principal Investigator — Västra Götalandsregionen
Locations (1):
- Västra Götalandsregionen, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No